CLINICAL TRIAL: NCT05397444
Title: Handgrip Strength (HGS) With HGS Asymmetry is Associated With All-cause Mortality and Hospital Readmissions Among Elderly Patients With Gastric Cancer.
Brief Title: Handgrip Strength (HGS) With HGS Asymmetry Are Associated With All-cause Mortality and Hospital Readmissions
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xueyi Miao, Principal Investigator, Nanjing Medical University
Other Study IDs: HGS ASYMMETRY
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Not
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Full robust: no low HGS without HGS asymmetry
  Interventions: Other: No intervention
- low HGS alone: low HGS without HGS asymmetry
  Interventions: Other: No intervention
- HGS asymmetry alone: no low HGS with HGS asymmetry
  Interventions: Other: No intervention
- low HGS with HGS asymmetry: non
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study with no intervention.

SUMMARY:
Adding the handgrip strength (HGS) asymmetry to the existing measurements of low HGS may improve the assessment of muscle function.

DETAILED DESCRIPTION:
We sought to explore the associations between maximal HGS with HGS asymmetry and mortality, hospital readmissions, total complications, and prolonged length of stay (PLOS) among elderly patients with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* with gastric cancer
* aged ≥60 years
* were scheduled to undergo radical surgery for the first time

Exclusion Criteria:

* received preoperative radiotherapy or chemotherapy
* combined with other types of malignant tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: elderly patients with gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | about 3 months
  within 3 months after surgery, collected from telephone follow-up
Hospital readmissions | about 3 months
  wihthin 3 months after surgery, collected from telephone follow-up

SECONDARY OUTCOMES:
Total complications | about 3 months
  during hospitalization, collected from medical records
prolonged length of stay | about 3 months
  during hospitalization, collected from medical records

CONTACTS AND LOCATIONS:
Overall Officials: xueyi miao, Principal Investigator — Nanjing Medical University
Locations (1):
- Nanjing medical university, Nanjing, China

IPD SHARING:
Plan to Share IPD: No